CLINICAL TRIAL: NCT00819208
Title: A Phase III Study of the Impact of a Physical Activity Program on Disease-Free Survival in Patients With High-Risk Stage II or Stage III Colon Cancer: A Randomized Controlled Trial
Brief Title: Health Education Materials With/Out a Physical Activity Program for Patients Who Have Undergone Treatment for High-Risk Stage II or Stage III Colon Cancer
Acronym: CHALLENGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Survivorship Research Group (Unknown); Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CO21; CAN-NCIC-CO21 (Registry Identifier: NCI US - Physician Data Query); CDR0000629834 (Other: PDQ)
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-02

CONDITIONS: Anxiety Disorder; Cognitive/Functional Effects; Colorectal Cancer; Depression; Fatigue; Psychosocial Effects of Cancer and Its Treatment; Sleep Disorders; Excercise
Keywords: fatigue; sleep disorders; depression; anxiety disorder; psychosocial effects of cancer and its treatment; cognitive/functional effects; stage II colon cancer; stage III colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Anxiety Disorders; Colorectal Neoplasms; Depression; Fatigue; Sleep Wake Disorders; Colonic Neoplasms | interventions — Counseling; Early Intervention, Educational; Therapeutics; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Program + General Health Education Materials (Active Comparator): Intervention Arm
  Interventions: Behavioral: exercise intervention; Other: counseling intervention; Other: educational intervention; Other: laboratory biomarker analysis; Other: questionnaire administration; Other: study of socioeconomic and demographic variables; Procedure: fatigue assessment and management; Procedure: quality-of-life assessment; Other: Fitness testing
- General Health Education Materials (Active Comparator): Control Arm
  Interventions: Other: laboratory biomarker analysis; Other: questionnaire administration; Other: study of socioeconomic and demographic variables; Procedure: fatigue assessment and management; Procedure: quality-of-life assessment; Other: Educational Intervention; Other: Fitness testing

INTERVENTIONS:
Behavioral: exercise intervention — 3 phases Phase 1: Intensive intervention for 6 months Phase 2: Reduced intervention for months 6-12 Phase 3: Minimal intervention for months 12-36
  Arms: Physical Activity Program + General Health Education Materials
Other: counseling intervention — Achieving an increase in PA from baseline of ≥ 10 MET hours/week will require a significant amount of behavioural support. The intervention will comprise a 36-month individualized PA and behavioural support program with a PAC. This will include a personalized PA prescription which takes into account the baseline fitness test results, PA history, performance status and patient's personal PA preferences and any barriers to activity. Most patients are likely to choose a walking program however any PA of at least moderate intensity level is acceptable.
  Arms: Physical Activity Program + General Health Education Materials
Other: educational intervention — Once at the beginning of the program
  Arms: Physical Activity Program + General Health Education Materials
Other: laboratory biomarker analysis — Every 12 months
Other: questionnaire administration — Every 6 months
Other: study of socioeconomic and demographic variables — Every 6 months
Procedure: fatigue assessment and management — Every 6 months
Procedure: quality-of-life assessment — Every 6 months
Other: Educational Intervention — For Arm 2 just once at beginning of program.
  Arms: General Health Education Materials
Other: Fitness testing — Objective fitness testing for both arms

SUMMARY:
RATIONALE: Participating in a physical activity program designed to increase free time physical activity and receiving written health education materials may influence the chance of cancer recurring as well as impact on physical fitness, psychological well-being and the quality of life of patients who have undergone surgery and chemotherapy for colon cancer. It is not yet known whether giving a physical activity program together with health education materials is more effective than giving health education materials alone for patients who have undergone colon cancer treatment.

PURPOSE: This randomized phase III trial is studying a physical activity program given together with health education materials to see how well it works compared with giving health education materials alone for patients who have undergone treatment for high-risk stage II or stage III colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the disease-free survival (DFS) of medically fit patients who have completed surgical resection and adjuvant chemotherapy for high-risk stage II or stage III colon cancer when administered a physical activity program with general health education materials vs general health education materials alone.

Secondary

* To compare the two intervention arms with respect to overall survival (OS); patient-reported outcomes using the SF-36, FACIT-F, PSQI, and HADS questionnaires; objective markers of physical fitness using body mass index, hip and waist circumference, submaximal exercise testing, and the Seniors' Fitness Test; physical activity behavior using the Total Physical Activity Questionnaire (TPAQ); safety profile as assessed by NCI CTCAE version 3.0; serum levels of insulin (i.e., IGF-1, IGF-2, and IGFBP3); cytokine levels (i.e., IL-1β, IL-6, IL-2, IL-4, IL-8, IL-10, IL-12, TNF-α, IFN-γ, and GM-CSF) and C-reactive protein levels; economic evaluations including cost-effective and cost-utility analyses; and predictors of physical activity adherence using the Social-Cognitive Determinants of Exercise Measure questionnaire.
* To evaluate the potential prognostic associations of the serum levels of insulin, IGF-1, IGF-2, IGFBP3, blood glucose, cytokines (i.e., IL- 1β, IL-6, IL-2, IL-4, IL-8, IL-10, IL-12, TNF-α, IFN-γ, and GM-CSF), and C-reactive protein with DFS, OS, level of physical activity, and level of fatigue in these patients.
* To evaluate the potential prognostic associations of age, gender, country, incremental increase in physical activity, and change in cardiovascular fitness with DFS, OS, level of fatigue, and quality of life in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to disease stage (II vs III), participating center, body mass index (≤ 27.5 vs > 27.5), and ECOG performance status (0 vs 1). Patients are randomized to 1 of 2 treatment interventions.

* Arm I: Patients receive general health education materials regarding nutrition and physical activity and undergo the Colon Health And Life Long Exercise Change (CHALLENGE) physical activity program consisting of behavior-support sessions and supervised physical activity sessions with a physical activity consultant.

  * Part I (intensive intervention for 6 months): Patients undergo 12 mandatory biweekly face-to-face behavior support sessions combined with 12 mandatory supervised physical activity sessions to increase their physical activity goal by 10 metabolic equivalent task (MET) hours/week. Twelve supervised physical activity sessions are also recommended on alternate weeks.
  * Part II (reduced intervention for months 6-12): Patients undergo 12 mandatory biweekly face-to-face or telephone behavior support sessions combined with 12 recommended supervised physical activity sessions to increase their physical activity goal by 20 MET hours/week.
  * Part III (minimal intervention for months 12-36): Patients undergo mandatory monthly face-to-face or telephone behavior support sessions combined with recommended supervised physical activity sessions to increase their physical activity goal to a maximum total of 27 MET hours/week.
* Arm II: Patients receive general health education materials regarding nutrition and physical activity.

Patients complete the Total Physical Activity Questionnaire (TPAQ) to assess exercise participation and undergo fitness testing periodically by the submaximal exercise test and Seniors' Fitness Test (SFT).

Patients complete the SF-36, FACT-F, Pittsburgh Sleep Quality Index (PSQI), Hospital Anxiety and Depression Scale (HADS), and Social Cognitive Determinants of Exercise Measure questionnaires periodically. Patients also complete a 30-day resource use diary and undergo a health economics analysis by the Work Productivity and Activity Impairment (WPAI) questionnaire.

Blood samples are collected periodically for correlative studies and fasting glucose. Samples are analyzed for markers of insulin level, IGF-1, IGF-2, and IGFBP3, cytokine levels (i.e., IL-1β, IL-6, IL-2, IL-4, IL-8, IL-10, IL-12, TNF-α, IFN-γ, and GM-CSF), and C-reactive protein levels.

During the 3 year intervention period, patients are followed every 6 months for 3 years and then annually for 4-10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Completely resected histologically confirmed adenocarcinoma of the colon

  * High-risk stage II disease, including one of the following:

    * T4 lesions
    * Less than 12 sampled lymph nodes
    * Poorly differentiated histology
  * Stage III disease, defined as having at least one pathologically confirmed positive lymph node or one pathologically confirmed positive tumour deposit.
  * Synchronous primary colon cancer allowed
* Adjuvant chemotherapy treatment for colon cancer with a 5-fluorouracil- based regimen received with an intent to provide a complete course of treatment. While one current standard is 24 weeks of treatment, patients who are pre-planned to receive a shorter duration of chemotherapy, including as part of a research study will also be permitted. The actual treatment received may be less than 24 weeks; participants must have received a minimum of one treatment cycle.
* Chemotherapy must have been completed (i.e. last dose received) a minimum of 60 days and a maximum of 180 days prior to registration.
* Carcinoembryonic antigen (CEA) ≤ 5 μg/L
* Current physical activity levels do not meet the recommended guidelines (≥ 150 minutes of moderate-to-vigorous or ≥ 75 minutes of vigorous physical activity/week) as calculated using the Leisure Time Exercise Questionnaire (LTEQ)
* Completion of chest x-ray or CT, and CT, MRI or ultrasound of abdomen within 60 days of registration; these imaging tests must not show evidence of metastatic or locally-recurrent colon cancer.
* Complete one of the following: (a) at least 2 stages of the submaximal exercise test with an acceptable heart rate and blood pressure response as defined in Appendix XII or (b) the 6 minute walk test with an acceptable heart rate and blood pressure response
* No rectal cancer

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Absolute granulocyte count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 100 g/L
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 times ULN
* ALT < 2 times ULN
* Not pregnant or planning to become pregnant within the next 3 years
* Able (i.e., sufficiently fluent) and willing to effectively communicate with the physical activity consultant affiliated with the originating cancer center
* Able (i.e., sufficiently fluent in English or French) and willing to complete the patient-reported outcome questionnaires, social determinants of exercise measurement, health economics, and physical activity questionnaires and logs
* Able to complete the baseline exercise test
* No significant comorbid conditions precluding participation in a physical activity program as determined by the investigator
* Likely to participate in a physical activity program, as assessed by the investigator
* No history of other malignancies, except adequately treated nonmelanoma skin cancer, curatively treated in situ cancer of the cervix, other solid tumors, Hodgkin lymphoma, or non-Hodgkin lymphoma curatively treated with no evidence of disease for > 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy as a component of treatment for primary tumor
* No concurrent treatment with additional chemotherapy or radiation
* No concurrent treatment with any medications deemed by the investigator as likely to preclude participation in a physical activity program
* No concurrent anticancer treatment including chemotherapy, biological, or targeted agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 889 (Actual)
Dates: Start 2009-06-02 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 10 years

SECONDARY OUTCOMES:
Overall survival | 10 years
Patient-reported outcomes, including quality of life, using SF-36, FACIT-F, PSQI, and HADS questionnaires | 5 years
Objective markers of physical fitness (i.e., body mass index, hip and waist circumference, cardiovascular fitness, and physical function) | 3 years
Physical activity behavior as assessed by TPAQ | 5 years
Safety profile according to NCI CTCAE version 3.0 | 10 years
Correlative biological markers including biochemical and molecular markers associated with insulin-related growth factor and cytokines associated with the mechanisms of fatigue | 3 years
Economic evaluations including cost-effective analysis and cost utility analysis | 5 years
Predictors of physical activity adherence as assessed by Social Cognitive Determinants of Exercise questionnaire | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Courneya, PhD, Study Chair — University of Alberta; Christopher Booth, MD, Study Chair — Cancer Centre of Southeastern Ontario at Kingston General Hospital; Janette Vardy, PhD, FRACP, Study Chair — Sydney Cancer Centre at Concord Repatriation General Hospital
Locations (47):
- United States (3):
  - Henry Ford Hospital, Detroit, Michigan
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- Australia (20):
  - Armidale Hospital, Armidale, New South Wales
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - North Coast Cancer Institute Coffs Harbour, Coffs Harbour, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Newcastle Private Hospital, Newcastle, New South Wales
  - North Coast Cancer Institute - Port Macquarie, Port Macquarie, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Tamworth Hospital, Tamworth, New South Wales
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandra, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Macarthur Cancer Therapy Centre - Campbelltown Hospital, Campbelltown
- Canada (21):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Horizon Health Network, Fredericton, New Brunswick
  - The Moncton Hospital, Moncton, New Brunswick
  - Regional Health Authority B, Zone 2, Saint John, New Brunswick
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Toronto Rehab, Toronto, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Sinai Health System, Toronto, Ontario
  - Lévis, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Montpellier, France
- Exercise Medicine Center for Diabetes and Cancer, Seoul, South Korea
- Belfast City Hospital, Belfast, Co. Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Courneya KS, Booth CM, Gill S, O'Brien P, Vardy J, Friedenreich CM, Au HJ, Brundage MD, Tu D, Dhillon H, Meyer RM. The Colon Health and Life-Long Exercise Change trial: a randomized trial of the National Cancer Institute of Canada Clinical Trials Group. Curr Oncol. 2008 Dec;15(6):279-85. doi: 10.3747/co.v15i6.378. PMID 19079628
- [Background] Vallance J, Lesniak SL, Belanger LJ, Courneya KS. Development and assessment of a physical activity guidebook for the Colon Health and Life-Long Exercise Change (CHALLENGE) trial (NCIC CO.21). J Phys Act Health. 2010 Nov;7(6):794-801. doi: 10.1123/jpah.7.6.794. PMID 21088311
- [Result] Courneya KS, Vardy JL, O'Callaghan CJ, Friedenreich CM, Campbell KL, Prapavessis H, Crawford JJ, O'Brien P, Dhillon HM, Jonker DJ, Chua NS, Lupichuk S, Sanatani MS, Gill S, Meyer RM, Begbie S, Bonaventura T, Burge ME, Turner J, Tu D, Booth CM. Effects of a Structured Exercise Program on Physical Activity and Fitness in Colon Cancer Survivors: One Year Feasibility Results from the CHALLENGE Trial. Cancer Epidemiol Biomarkers Prev. 2016 Jun;25(6):969-77. doi: 10.1158/1055-9965.EPI-15-1267. Epub 2016 Apr 8. PMID 27197271
- [Derived] Courneya KS, Booth CM, Vardy JL, Friedenreich CM, Dhillon HM, Coyle V, Campbell KL, Arthuso FZ, Turner J, Kent DE, Russell C, Gordon JJ, Henson J, Chua NS, Jonker DJ, Kay S, Gill S, O'Brien P, Tu D, O'Callaghan CJ. Effects of a structured exercise program on motivational outcomes in patients with Colon cancer. J Natl Cancer Inst. 2026 Jan 29:djag023. doi: 10.1093/jnci/djag023. Online ahead of print. PMID 41609410
- [Derived] Courneya KS, Vardy JL, O'Callaghan CJ, Gill S, Friedenreich CM, Wong RKS, Dhillon HM, Coyle V, Chua NS, Jonker DJ, Beale PJ, Haider K, Tang PA, Bonaventura T, Wong R, Lim HJ, Burge ME, Hubay S, Sanatani M, Campbell KL, Arthuso FZ, Turner J, Meyer RM, Brundage M, O'Brien P, Tu D, Booth CM; CHALLENGE Investigators. Structured Exercise after Adjuvant Chemotherapy for Colon Cancer. N Engl J Med. 2025 Jul 3;393(1):13-25. doi: 10.1056/NEJMoa2502760. Epub 2025 Jun 1. PMID 40450658